CLINICAL TRIAL: NCT01284777
Title: Nuclear Matrix and Cancer: Proteomic and Genomic Analyses Using Microarray in Cells Obtained Via Thoracocentesis
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-A00295-34; 2010-01 (Other: internal number)
Record Dates: First submitted 2010-05-18; First posted 2011-01-27 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Cancer
Keywords: cancerology; genetic
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection; Thoracentesis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients
  Interventions: Genetic: blood sample, thoracocentesis

INTERVENTIONS:
Genetic: blood sample, thoracocentesis — 20ml of blood only one thoracocentesis (the same that one for diagnostic)

SUMMARY:
Accurate characterization of malignant cells obtained via thoracocentesis is of paramount importance in the management of cancer patients. The identification of novel biomarkers may in that regard considerably improve the diagnostic approach of these pleural effusions, guide therapeutic decisions, particularly with respect to targeted therapies, and offer helpful prognostic information. Nuclear anomalies represent the cornerstone of the cytologic and/or histopathologic diagnosis of malignant cells. The nuclear matrix is a fundamental constituent of the nuclear architecture via its interaction with the nuclear membrane, but is also directly involved with DNA and RNA processing. Prior studies have suggested that in some cancers, the lamins, a major constituent of the nuclear matrix, have different patterns of expression or nuclear localization that could potentially have prognostic implications. Our project aims at studying the constituents of the nuclear matrix of malignant cells isolated for pleural fluid in patients with metastatic disease, both of bronchogenic or non-bronchogenic origin, which, to our knowledge, has not yet been done. Both proteomic (localization by immunofluorescence and expression by Western-Blot) and genomic (microarray, CGH type) analyses will be undertaken to identify microrearrangements in the genes of interest. The primary aim is to identify specific biomarkers to more accurately characterize malignant cells in metastatic pleural disease.

ELIGIBILITY:
Inclusion Criteria:

* sign consent approval
* patients with metastatic disease, both of bronchogenic or non-bronchogenic origin
* 50% or more of malignant cells

Exclusion Criteria:

* patients with tumoral treatment during thoracocentesis
* 50% or less of malignant cells

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with metastatic disease
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
identify specific biomarkers to more accurately characterize malignant cells in metastatic pleural disease | 2 years
  Research for quantitative or qualitative nuclear-matrix-proteins anomalies in secondary metastatic pleural disease and/or for anomalies in the genes coding for these proteins.
  Protein analysis : immunofluorenscy, western blot. Genomic analysis : CGH arrays.

SECONDARY OUTCOMES:
Variations of nuclear matrix proteins expression or localization in malignant cells released in pleural liquid | 2 years
Comparison of nuclear matrix protein expression in metastatic cells | 2 years
  by taking account of the origin and the histological nature of the primitive tumor
Identify genomic anomalies of the interest genes | 2 years
  the tumoral cells genome versus the peripheral cells genome
Search existence of a correlation between the quantity of expressed proteins and the number of genes copies in the tumoral cells | 2 years
Compare their results with the data published on cell-lineages and on tissular samples | 2 years
  Showing differences between tumor cells, cell-lineages and cells released in the liquid

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Roll, Principal Investigator — Assistance Publique des Hôpitaux de Marseille
Locations (2):
- France (2):
  - Assistance Publique des Hôpitaux de Marseille, Marseille
  - Assistance Publique Hopitaux de Marseille, Marseille